CLINICAL TRIAL: NCT04149067
Title: Retrospective and Multicenter Study of Real-world Evidence With SGLT2i (Dapagliflozin) and DPP4i (Sitagliptin) in Type 2 Diabetes Patients in Spain
Brief Title: Study of Real-world Evidence With SGLT2i (Dapagliflozin) and DPP4i (Sitagliptin) in Type 2 Diabetes Patients in Spain
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: FIS-DAP-2016-01
Record Dates: First submitted 2019-09-17; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dapagliflozin cohort: Patients diagnosed with type 2 diabetes that started dapagliflozin treatment at least 6 months before the beginning of the study.
  Interventions: Drug: Dapagliflozin
- Sitagliptin cohort: Patients diagnosed with type 2 diabetes that started sitagliptin treatment at least 6 months before the beginning of the study.
  Interventions: Drug: Sitagliptin

INTERVENTIONS:
Drug: Dapagliflozin — Evaluation of the effectiveness and safety of the Dapagliflozin treatment.
  Other Names: iSGLT2
  Groups: Dapagliflozin cohort
Drug: Sitagliptin — Evaluation of the effectiveness and safety of the Sitagliptin treatment.
  Other Names: iDPP4
  Groups: Sitagliptin cohort

SUMMARY:
The aim of this study is to develop a retrospective, multicenter and observational study in Spain in real clinical practice to assess the employment of dapagliflozin and to compare its effectiveness and safety with the data of sitagliptin, a DPP4 inhibitor. This is a widely used molecule in Spain with a large safety profile. It was chosen as a comparator because of the number of patients treated and because it is a real alternative at the time of making a decision about the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with T2DM.
2. Age: 18-75 years.
3. Treatment with dapagliflozin or sitagliptin that started at least 6 months before the recruitment date.
4. The patient must have at least two follow-up visits. The basal initial visit, where all the relevant information is collected and a second follow-up visit.
5. The next information of the subjects should be available at the recruitment of the basal visit: Sex, age (years), date of diagnosis of T2DM, weight, height, systolic and diastolic blood pressure, body mass index (BMI: kg / m2), concomitant medication (antiHTA, statins, aspirin, etc.), glucose basal fasting (mg / dL), HbA1c (%) and estimated GFR by CKD-EPI (mL / min / 1.73m2).

5. The patient must sign the informed consent to participate in the study.

Exclusion Criteria:

1. Impediment of the patient to give him informed consent.
2. Patients diagnosed with Type 1 Diabetes.
3. Women with gestational diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old with stable DM2 with antihyperglycaemic therapy, being included in their treatment dapagliflozin or sitagliptin medication.
Sampling Method: Non-Probability Sample
Enrollment: 1080 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
0.5% in Hb1Ac and 1.5 kg in body weight | 6 months +/- 3 months
  The aim of the study is to assess the effectiveness of the SGLT2i (dapagliflozin) and DPP4i (Sitagliptin) over the composite endpoint of Hb1Ac and weight at six month of treatment.
  The main variable is composite, including Hb1Ac and body weight. It will be evaluated the proportion of patient to achieve a change of 0.5% in Hb1Ac and 1.5 kg in body weight.
  It was chosen sitagliptin because the researchers involved in this study have much experience with this molecule with a large number of patients already treated.

SECONDARY OUTCOMES:
Evaluate the results due to the use of SGLT2i/DPP4i | 6 months +/- 3 months
  Assessment of the SGLT2i/DPP4i use in single, double or triple therapy and analysis of the baseline features of the patients at the beginning and at the end of the treatment, including the concomitant medication.
Evaluate the security of the treatment | 6 months +/- 3 months
  Study of the incidence of the urinary and genital infections as well as the hypoglycemia incidence and its severity.

CONTACTS AND LOCATIONS:
Overall Officials: Cristobal Morales Portillo, Study Director — Hospital Universitario Virgen Macarena
Locations (1):
- Cristóbal Morales Portillo, Seville, Andalusia, Spain